CLINICAL TRIAL: NCT07252882
Title: Interest of Magnetic Resonance Imaging in the Diagnosis of Upper Urinary Tract Invasive Tumours
Acronym: UUTICaD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/23/0389
Record Dates: First submitted 2025-06-20; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Magnetic Resonance Imaging (MRI); Urologic Cancer
Keywords: Upper urinary tract magnetic resonance imaging
MeSH Terms: conditions — Urologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with upper urinary tract tumour (Experimental): Patients with upper urinary tract tumour and will have upper urinary tract magnetic resonance imaging
  Interventions: Radiation: Upper urinary tract magnetic resonance imaging

INTERVENTIONS:
Radiation: Upper urinary tract magnetic resonance imaging — Patients with a suspected malignant tumour of the upper urinary excretory tract based on the presence of a suspicious lesion on a uro-computed tomography scan will have a diagnostic magnetic resonance imaging of the urinary tract with Gadolinium-based contrast agents

SUMMARY:
Upper urinary tract invasive cancer magnetic resonance imaging diagnosis

DETAILED DESCRIPTION:
Urothelial tumours are the 6th most common cause of cancer in developed countries and occur throughout the urinary tract (urethra, bladder, ureter and pelvic cavities). Upper urinary tract tumours account for 5-10% of urothelial carcinomas. Nearly 60% of patients with upper urinary tract tumours are diagnosed as invasive (≥ T2). 90% of computed tomography lesions are tumour lesions. Currently, the diagnosis of upper urinary tract tumours is based on computed tomography with injection of nephrotoxic iodinated contrast medium (uro-computed tomography) and biopsies taken during ureteroscopy under general anaesthesia. Invasive tumours have a poor prognosis and patients with infiltrating tumours may benefit from neoadjuvant chemotherapy prior to nephroureterectomy (which may impair renal function). Uro-computed tomography cannot differentiate between invasive and non-invasive tumours and biopsies taken in the operating theatre during ureteroscopy under general anaesthesia are unreliable for staging and frequently underestimate the disease. The diagnosis of infiltrating tumours is most often made on nephro-ureterectomy specimens, making neoadjuvant treatment impossible. Recently, functional magnetic resonance imaging sequences (diffusion weighted imaging, apparent diffusion coefficient) highlighted the biophysical properties of the tissues such as cellular organisation, density and microcirculation and have thus made it possible to differentiate benign from malignant lesions by identifying the level of tissue involvement. Magnetic resonance imaging has become a real tool in the diagnosis of bladder tumours and can differentiate between infiltrating and non-infiltrating lesions.

The aim of this study is to make magnetic resonance imaging for each patient and compare results to pathological analysis (nephro-ureterectomy pathologic analysis or biopsy with 3 months Uro-computed tomography) to evaluate magnetic resonance imaging diagnosis capability for invasive tumour.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age with a suspected upper urinary tract tumour based on the presence of a suspicious lesion on a uro-computed tomography scan
* Have given free, informed and signed consent
* Be affiliated to a social security scheme

Exclusion Criteria:

* Renal failure not allowing the injection of iodinated contrast media (Glomerular filtration rate <30mL/min)
* Subject under legal protection (guardianship or curatorship)
* Pregnant or breastfeeding woman
* Person participating in another research study or having participated in a protocol with an exclusion period still in progress at inclusion
* Contraindication to magnetic resonance imaging (patient with non-magnetic resonance imaging compatible equipment, claustrophobia preventing magnetic resonance imaging)
* Acide gadoteric hypersensibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic validity (composite criteria sensitivity and specifcity) of a predefined magnetic resonance imaging sequence in the diagnosis of upper urinary tract invasive tumour | 3 months
  Diagnostic validity (sensitivity and specifcity) of a predefined magnetic resonance imaging sequence in the diagnosis of upper urinary tract invasive tumour (taking as reference the pathological analysis [gold standard] or biopsy with 3 months Uro-CT).

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Hôpital Pellegrin, Bordeaux, France
  - Hôpital Claude Huriez, Lille, France
  - Institut Paoli Calmettes, Marseille, France
  - Clinique Beau Soleil, Montpellier, France
  - Hôpital Lapeyronie, Montpellier, France
  - Hôpital Saint-Louis, Paris, France
  - Hôpital de la Pitié Salpêtrière, Paris, France
  - Hôpital Européen Georges Pompidou, Paris, France
  - Clinique La Croix du Sud, Quint-Fonsegrives, France
  - CHU de Toulouse, Toulouse, France
  - Clinique Pasteur, Toulouse, France

IPD SHARING:
Plan to Share IPD: No